CLINICAL TRIAL: NCT00134836
Title: Preventive Primary Care Outreach for High Risk Older Persons
Acronym: PPCO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Jenny Ploeg, McMaster University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: PHCTF G03-02795
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Preventive Primary Care Outreach — Nurse home visit at baseline, 6 months, 12 months, including comprehensive assessment using MDS HC, care planning, referral to appropriate services
  Other Names: nurse home visit

SUMMARY:
It is recognized that a significant proportion of seniors over 75 years of age are at risk of functional decline, and thus of institutionalization and death. The investigators at McMaster University Medical Centre, are conducting is a randomized controlled trial of a preventive primary care outreach (PPCO) service provided to high risk seniors living in the community. The goal of this service is to identify unrecognized problems and individuals at increased risk and to link individuals to care. This preventive primary care service is provided by nurse case managers. The investigators have recruited patients through their family physicians who work in primary care networks. The investigators are screening all seniors aged 75 and over within these practices. The sample includes seniors aged 75 and over who are identified to be at risk according to the Sherbrooke Postal Questionnaire. Patients are randomly allocated to intervention and control groups. A research assistant, who is blind to group allocation, will collect data from seniors at baseline, six months, and at the end of one year.

Outcome measures include health-related quality of life (quality adjusted life years [QALYs]), health and social service utilization and costs, mortality, institutionalization, functional status, and perceived health status.

Primary Hypothesis:

The intervention compared to usual care will result in higher health-related quality of life.

Secondary Hypotheses:

Compared to usual care, the PPCO intervention will result in:

* the same or lower costs associated with service utilization;
* less functional decline;
* reduced mortality;
* lower rates of institutionalization; and
* better self-rated health.

DETAILED DESCRIPTION:
Seniors consume a large proportion of health care resources in Canada. It is recognized that a significant proportion of seniors over 75 years of age are at risk of functional decline, and thus of institutionalization and death. A recent meta-analysis of nineteen studies of preventive primary care outreach interventions with older persons found that such interventions were associated with a significant reduction of mortality (Summary Odds Ratio [OR] 0.83, 95% confidence interval [CI] 0.75 to 0.91) and an increased likelihood of living in the community (OR 1.23, 95% CI 1.06 to 1.43). While four of the nineteen studies were conducted in Canada, none of these examined health-related quality of life or the cost effectiveness of the intervention.

The study we are conducting is a randomized controlled trial of a preventive primary care outreach service provided to high risk seniors living in the community. The goal of this service is to identify unrecognized problems and individuals at increased risk and to link individuals to care. This preventive primary care service is provided by nurse case managers. At an initial home visit, the nurse will conduct a comprehensive, multidimensional assessment, identify problems and develop a plan of care, using the Minimum Data Set for Home Care and Client Assessment Protocols. The nurse will work with the senior and the family physician to plan and implement care. While frequency of home and phone visits will depend on the needs of seniors, it is expected that, on average, seniors in the intervention group will receive 10 hours of nursing contact during the one year of intervention.

We have recruited primary care networks and family physician practices within these networks. Within these practices, we are screening all seniors aged 75 and over. The sample includes seniors aged 75 and over who are identified to be at risk according to the Sherbrooke Postal Questionnaire. We will recruit 640 patients for the study and randomly allocate them to intervention and control groups. A research assistant, who is blind to group allocation, will collect data from seniors at baseline, six months, and at the end of one year.

Outcome measures include health-related quality of life (quality adjusted life years [QALYs]), health and social service utilization and costs, mortality, institutionalization, functional status, and perceived health status.

Primary Hypothesis:

The intervention compared to usual care will result in higher health-related quality of life.

Secondary Hypotheses:

Compared to usual care, the PPCO intervention will result in:

* the same or lower costs associated with service utilization;
* less functional decline;
* reduced mortality;
* lower rates of institutionalization; and
* better self-rated health.

The available evidence regarding the effectiveness and economic impact of primary care interventions with seniors is inadequate for the development of health care policy in Ontario and Canada. The present proposal employs a research design that addresses the limitations of research conducted to date. The results of this study will guide policy makers in addressing problems in primary care for seniors and assist in decision making related to services for high risk seniors.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 75 years of age and older
* Patient is listed on the roster of a participating family physician practice
* Patient resides in the Hamilton, Ontario, Canada area
* Patient or proxy able to answer questions in English

Exclusion Criteria:

* Principal residence is nursing home or long term care facility
* Patient is identified by family physician as palliative
* Patient currently receives home care services through the Community Care Access Centre
* Patient is a 'snowbird' and out of town for more than four weeks in any year
* Patient is scheduled for major elective surgery in the next year

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 719 (Actual)
Dates: Start 2004-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (quality adjusted life years [QALYs]) | baseline, 6 months, 12 months

SECONDARY OUTCOMES:
Health and social service utilization and costs | baseline, 6 months, 12 months
mortality | 12 months
institutionalization | 12 months
functional status | baseline, 6 months, 12 months
perceived health status | baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Ploeg, RN, PhD, Principal Investigator — School of Nursing, Faculty of Health Sciences, McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Ploeg J, Brazil K, Hutchison B, Kaczorowski J, Dalby DM, Goldsmith CH, Furlong W. Effect of preventive primary care outreach on health related quality of life among older adults at risk of functional decline: randomised controlled trial. BMJ. 2010 Apr 16;340:c1480. doi: 10.1136/bmj.c1480. PMID 20400483